CLINICAL TRIAL: NCT05365802
Title: PET Study of 68Ga-FAPi-46 in Patients With Interstitial Lung Disease: an Exploratory Biodistribution Study With Histopathology Validation.
Brief Title: FAPI PET for Lung Fibrosis
Acronym: FAPI ILD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jeremie Calais, Clinical Research Director, Ahmanson Translational Theranostics, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB21-000678
Record Dates: First submitted 2022-04-22; First posted 2022-05-09 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Interstitial Lung Disease; Idiopathic Interstitial Pneumonias; Drug-Induced Pneumonitis; Hypersensitivity Pneumonitis; Radiation Pneumonitis; Pneumoconiosis; Pulmonary Fibrosis
Keywords: interstitial lung disease; pulmonary fibrosis; 68Ga-FAPi-46
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Interstitial Pneumonias; Alveolitis, Extrinsic Allergic; Radiation Pneumonitis; Pneumoconiosis; Pulmonary Fibrosis | interventions — FAPI-46; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 68Ga-FAPi-46 (Experimental): Patients receive 68Ga-FAPi-46 IV and undergo PET/CT scan over 20-50 minutes
  Interventions: Drug: 68Ga-FAPi-46; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: High Resolution Computed Tomography

INTERVENTIONS:
Drug: 68Ga-FAPi-46 — Radiopharmaceutical will be administered via IV
  Other Names: Gallium-68-FAPi-46
Procedure: Computed Tomography — As part of PET/CT scan
  Other Names: CT scan
Procedure: Positron Emission Tomography — As part of PET/CT scan
  Other Names: PET scan
Procedure: High Resolution Computed Tomography — Will be conducted immediately after FAPI PET/CT

SUMMARY:
This is a prospective exploratory biodistribution study in patients with interstitial lung disease (ILD).

The purpose of this research study is to determine where and to which degree the FAPI tracer (68Ga-FAPI-46) accumulates in normal and fibrotic lung tissues of patients with interstitial lung disease.

The study will include patients with interstitial lung disease who have or will initiate a new ILD medication OR will undergo tissue biopsy or surgery of the lung.

The study will include 30 patients, the upper limit for PET imaging studies conducted under the Radioactive Drug Research Committee (RDRC) purview.

Participants will be injected with up to 7 mCi of 68-GaFAPi and will undergo one PET/CT scan and one High Resolution CT of the lungs.

The study is sponsored by Ahmanson Translational Theranostic Division at UCLA.

DETAILED DESCRIPTION:
ILD is a group of respiratory diseases that affect the interstitium of the lungs. A major problem is the highly variable course of fibrosing ILD: some patients remain stable without treatment, and others progress rapidly despite pharmacotherapy.

Novel diagnostic approaches for risk stratification with more accurate prediction of the course of fibrosing ILD could potentially improve prognostication and ultimately lead to better survival in these patients.

Persistent activation and local accumulation of myofibroblasts is a common feature of fibrotic diseases. FAP is a promising target for molecular imaging of fibroblast activation and detection of sites of active tissue remodeling.

Small molecule inhibitors of FAP have been labeled with positron-emitting isotopes for PET imaging. 68Ga-FAPi-46 can serve as diagnostic biomarker in ILD.

In this study, the investigators will evaluate the 68Ga-FAPi-46 biodistribution in patients with ILD and observe the correlation of FAP expression and FAPi radiopharmaceutical uptake.

The primary objective of this study is to evaluate the biodistribution of the new FAP-targeted PET tracer, 68Ga-FAPi- 46, in patients with ILD.

OUTLINE:

1. Participants with Interstitial Lung Disease will be asked to undergo a 68Ga-FAPi-46 PET/CT and one High Resolution CT of the lungs
2. Patients will be followed until pathology is obtained during clinical care. (if undergoing surgery or biopsy)
3. Biodistribution results will be assessed comparing pathological findings and PET/CT results

ELIGIBILITY:
Inclusion criteria

* Patients with ILD confirmed by CT at time of staging
* Patients who have initiated or will initiate a new ILD medication with 3 months of enrollment OR Patients who are scheduled to undergo tissue biopsy or surgery of the lung
* Patients are ≥ 18 years old at the time of the radiotracer administration
* Patient can provide written informed consent

Exclusion criteria

* Patient is pregnant or nursing
* Patients with active infectious lung disease
* Patients not expected to comply with the protocol requirements, not able to understand or follow trial procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To define and document the biodistribution of gallium Ga 68 FAPi-46 (68Ga-FAPi-46) in patients with Interstitial Lung Disease | 60 minutes following injection
  To quantify diseased tissue and normal background organs, 68Ga-FAPI-46 positron emission tomography (PET) tracer biodistribution will be assessed by semi-quantitative analysis (unit/metrics = standardized uptake values (SUV)).

SECONDARY OUTCOMES:
68Ga-FAPi-46 accumulation | Up to 2 years
  To evaluate the degree of 68Ga-FAPi-46 accumulation observed by PET imaging as opposed to the amount of FAP expression in obtained lung tissue, when available. IHC will be scored with a semi-quantitative scoring system that accounts for staining intensity (0-2, where 0 is negative, 1 is weak, 2 is strong and eq. stands for equivocal). Correlations will be sought using least square regression analysis.
68Ga-FAPi-46 and disease progression | Up to 2 years
  To evaluate whether the 68Ga-FAPi-46 biodistribution in the lungs can be associated with disease progression under ILD therapies.
68Ga-FAPi-46 biodistribution | Up to 2 years
  To evaluate whether the 68Ga-FAPi-46 biodistribution in the lungs can be associated with HR CT quantitative parameters

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, MD, Principal Investigator — Clinical Research Director, Ahmanson Translational Theranostics
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No